CLINICAL TRIAL: NCT02562664
Title: Insulin Sensitizing Agent (Metformin) Improves Clinical Pregnancy Rate and Insulin Parameters in Polycystic Ovarian Syndrome Patients With Acanthosis Nigricans
Brief Title: Metformin Improves Clinical Pregnancy Rate in Polycystic Ovarian Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPCOS
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Reproductive Endocrinology; Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CC with placebo (Active Comparator): 100 mg clomiphene Citrate (Clomid , global Napi , Egypt) CC tablets taken from day 3 to day 7 of the cycle with placebo tablets taken twice daily continuously for three cycles.
  Interventions: Drug: CC; Drug: Placebo tablets
- CC plus Metformin (Active Comparator): received t100 mg clomiphene Citrate (Clomid , global Napi , Egypt) CC tablets taken from day 3 to day 7 of the cycle with plus Metformin 500 mg twice daily continuously for three cycles.
  Interventions: Drug: CC; Drug: Metformin

INTERVENTIONS:
Drug: CC — 100 mg clomiphene Citrate (Clomid , global Napi , Egypt) CC tablets taken from day 3 to day 7 of the cycle
Drug: Placebo tablets — Placebo tablets taken twice daily continuously for three cycles.
  Arms: CC with placebo
Drug: Metformin — wMetformin (Cidophage , Amon , Egypt) 500 mg twice daily continuously for three cycles.
  Arms: CC plus Metformin

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common Female endocrine disorder , with a prevalence ranging between 6% to10% based on the National Institutes of Health (NIH) criteria and when the broader Rotterdam criteria are applied it reaches as high as 15%. Typically, PCOS can identify during the early adolescence. Insulin resistance is a common finding in the obese women with PCOS. It is most prevalent and severe in PCOS phenotype involving hyperandrogenism and chronic anovulation. Women with PCOS who have regular cycles are metabolically less abnormal. Acanthosis nigricans (AN) is a dermatosis characterized by velvety, papillomatous, brownish-black, hyperkeratotic plaques, typically of the intertriginous surfaces and neck. Although AN is associated with malignancy, the recognition of its more common connection to obesity and insulin resistance allows for diagnosis of related disorders including type 2 diabetes, the metabolic syndrome, and polycystic ovary syndrome. Significant improvements in ovulation and pregnancy rates as a result of clomiphene treatment after metformin in women with clomiphene-resistant PCOS were reported in a popular randomized, double-blind, placebo-controlled trial . The first pharmacological approach to induction of ovulation in women with PCOS is clomiphene citrate

ELIGIBILITY:
Inclusion Criteria:

* All patients with PCOS fulfilled at least 2 out of the three criteria of Rotterdam consensus 2003

Exclusion Criteria:

* liver disease
* heart or respiratory failure
* alcohol abuse
* kidney disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 6 months

SECONDARY OUTCOMES:
Fasting glucose (mg/dl) | 6 months
Fasting insulin (mg/dl) | 6 months